CLINICAL TRIAL: NCT02465710
Title: Comparisons of Clinical Outcomes Between Novel Tailored Transvaginal Mesh Surgery and Vaginal Native Tissue Repair Surgery for Pelvic Organ Prolapse
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201504023RINC
Record Dates: First submitted 2015-06-04; First posted 2015-06-08 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Pelvic Organ Prolapse
Keywords: pelvic organ prolapse; pelvic floor reconstruction surgery; transvaginal mesh surgery; Women; Surgical treatment
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Melanocyte-Stimulating Hormones

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- pelvic organ prolapse: All women who underwent surgical treatment of pelvic organ prolapse in this study.
  Interventions: Procedure: Pelvic organ prolapse surgery without mesh; Procedure: Pelvic organ prolapse surgery with mesh

INTERVENTIONS:
Procedure: Pelvic organ prolapse surgery without mesh — retrospective study
Procedure: Pelvic organ prolapse surgery with mesh

SUMMARY:
The issue of whether utilizing the mesh in the surgical treatment of pelvic organ prolapse remained undetermined.Thus, the aim of this study is to analyze clinical outcome of women who underwent pelvic organ prolapse surgeries with and without mesh implantation in the Department of Obstetrics & Gynecology of National Taiwan University Hospital.

DETAILED DESCRIPTION:
Hypothesis / aims of study:

The use of mesh for women with pelvic organ prolapsed (POP) remains under debate, despite a recent randomized trial reported a favourable anatomic outcome of transvaginal mesh (TVM) surgery for cystocele, compared with anterior colporrhaphy. Besides, the issue of preserving uterus or not in women with POP during operation is still undetermined. Thus, the aim of this study is to compare clinical outcomes of the novel tailored TVM surgeries and conventional transvaginal native tissue repair (NTR) surgeries for POP.

Study design, materials and methods:

Between November 2011 and September 2014, the medical records of all consecutive women who underwent POP surgeries in a medical centre were reviewed. The choice of surgery method was according to the surgeons' preference. Clinical characteristics and intraoperative data and postoperative clinical outcomes were recorded. Wilcoxon rank-sum test was used to compare the data between two groups. Kaplan-Meier survival analysis was used to compare the recurrence rate between two groups.

ELIGIBILITY:
Inclusion Criteria:

* All women who underwent surgical treatment of pelvic organ prolapse were enrolled in this study.
* ≥ 20 years old female.

Exclusion Criteria:

* Healthy women
* Without underwent surgical treatment of pelvic organ prolapse

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All women who underwent surgical treatment of pelvic organ prolapse were enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate of pelvic organ prolapse | 5 years
  follow-up till postoperative 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics & Gynecology, National Taiwan University Hospital, Taipei, Taiwan, Taiwan